CLINICAL TRIAL: NCT05941715
Title: Faricimab for High-frequent Aflibercept Treated Neovascular Age-related Macular Degeneration: a Monocenter, Randomized, Double-masked Comparator-controlled Study (FAN)
Brief Title: Faricimab for High-frequent Aflibercept Treated Neovascular Age-related Macular Degeneration
Acronym: FAN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 35-200 ex 22/23; 2023-000037-32 (EudraCT Number)
Record Dates: First submitted 2023-06-19; First posted 2023-07-12 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: aflibercept; faricimab; treat and extend; nAMD; AMD; neovascular age-related macular degeneration
MeSH Terms: interventions — aflibercept; faricimab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group A: aflibercept first (part 1), switch to faricimab (part 2) (Active Comparator): Aflibercept 2.0mg/0.05ml intravitreal will be administered from baseline through to the first visit at or after 32 weeks in a treat-and-extend regime.
  At the first visit at or after 32 weeks, faricimab 6.0mg/0.05ml intravitreal will be administered in a treat-and-extend regime through to the last visit before 56 weeks.
  Interventions: Drug: Aflibercept 40 MG/ML; Drug: Faricimab 120 MG/ML
- group B: faricimab monotherapy (Experimental): Faricimab 6.0mg/0.05ml intravitreal will be administered from baseline through to the last visit before 56 weeks in a treat-and-extend regime.
  Interventions: Drug: Faricimab 120 MG/ML

INTERVENTIONS:
Drug: Aflibercept 40 MG/ML — treat-and-extend
  Other Names: Eylea®
  Arms: group A: aflibercept first (part 1), switch to faricimab (part 2)
Drug: Faricimab 120 MG/ML — treat-and-extend
  Other Names: Vabysmo®

SUMMARY:
Study purpose: To evaluate if previously high-frequent (3-5 weekly) aflibercept treated neovascular age-related macular degeneration (nAMD) can be extended in their treatment interval when switched to faricimab.

Primary objective: To assess the efficacy of faricimab compared to aflibercept in terms of durability at 32 weeks by extending treatment interval in previous high-frequent aflibercept treated nAMD.

DETAILED DESCRIPTION:
There is a subgroup of nAMD patient requiring monthly interventions, when applying as needed and treat-and-extend treatment strategies. A burden for both patient/caregivers and health care systems. More durable treatment options are needed to increase the quality of life for these nAMD patients, as well as to make human resources available for the growing elderly AMD population requiring treatment.

The FAN study is a randomized, double-masked, 2-arm (comparator-controlled), phase-IV, monocenter study with a primary endpoint at 32 weeks. The study is conducted into 2 parts. Patients will receive either aflibercept or faricimab via treat-and-extend principle until the primary endpoint (part 1). As mentioned, the main objective is to assess the durability of both drugs in this particular subgroup of nAMD patients. In part 2 of the study, starting at or after 32 weeks, all patients will receive faricimab via treat-and-extend until the end of the study (56 weeks).

ELIGIBILITY:
Ocular inclusion criteria:

* MNV due to AMD (nAMD)
* BVCA between and including 19 and 75 letters (Snellen equivalent approximately 20/400 to 20/32)
* ≥ 7 previous intravitreal injections with anti-VEGF
* the last ≥ 4 consecutive intravitreal injections with aflibercept
* the last aflibercept injections within the last 35 days
* interval between the last 2 aflibercept injections ≤ 35 days

Ocular exclusion criteria:

* MNV due to other causes than nAMD
* polypoidal choroidal neovascularization
* retinal pigment epithelial rip/tear
* subretinal hemorrhage of > 50% of the lesion, involving the fovea
* any macular pathology other than AMD causing structural changes of the macula and thereby affecting vision
* any active intra-/periocular infection/inflammation of the study eye
* uncontrolled glaucoma under medication (IOP >25mmHg)
* cataract surgery of the study eye within the last 3 months
* previous intraocular surgery of the study eye other than cataract surgery or intravitreal injections with anti-VEGF (e.g. vitrectomy, corneal transplant, glaucoma surgery)
* any previous laser therapy of the study eye other than Yag (yttrium aluminium garnet) laser capsulotomy (e.g. panretinal photocoagulation, verteporfin photodynamic therapy)
* refractive error of more than -6 diopters myopia
* vitreous hemorrhage
* retinal detachment

General exclusion criteria

* use of long-term systemic corticosteroids within the last 3 months
* uncontrolled blood pressure (either/both systolic blood pressure >180mmHg, diastolic blood pressure >100mmHg)
* pregnancy (pre-menopausal women MUST take a pregnancy test at time of initiation)
* breast-feeding
* myocardial infarction or stroke within the last six months
* concomitant participation in another clinical study with investigational medicinal products
* a known allergy or hypersensitivity towards eye drops needed for the examinations planned during the study, and/or the intravitreal procedure.
* a known allergy or hypersensitivity against fluorescein / indocyanine green used during angiography
* a known allergy or hypersensitivity towards any of the components of the study drug

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-07-04 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2025-02-26 (Actual)

PRIMARY OUTCOMES:
Proportion of eyes with at least one extension without retinal (intra- and subretinal) fluid within the time period baseline to 32 weeks (extension success rate) | at 32 weeks
  Treatment is administered at each visit. The interval between treatments is based on a treat and extend regime. The first interval between treatments, from baseline, is 4 weeks. Intra- and subretinal fluid are assessed at each visit with optical coherence tomography (OCT). Should no intra- and subretinal fluid be present on OCT, the treatment interval to the next visit is extended by 2 weeks. Is intra- and or subretinal fluid present on OCT the treatment interval to the next visit is reduced by 2 weeks. The minimum treatment interval is 4 weeks, the maximum treatment interval is 12 weeks.

SECONDARY OUTCOMES:
Proportion of eyes with maximum extended interval without retinal (intra- and subretinal) fluid of ≥ 6, ≥ 8, ≥ 10 weeks and (≥ 12weeks) | at 32 weeks and 56 weeks
  Treatment is administered at each visit. The interval between treatments is based on a treat and extend regime. The first interval between treatments, from baseline, is 4 weeks. Intra- and subretinal fluid are assessed at each visit with optical coherence tomography (OCT). Should no intra- and subretinal fluid be present on OCT, the treatment interval to the next visit is extended by 2 weeks. Is intra- and or subretinal fluid present on OCT the treatment interval to the next visit is reduced by 2 weeks. The minimum treatment interval is 4 weeks, the maximum treatment interval is 12 weeks.
Maximum extended treatment interval without retinal (intra- and subretinal) fluid | at 32 weeks and 56 weeks
  Treatment is administered at each visit. The interval between treatments is based on a treat and extend regime. The first interval between treatments, from baseline, is 4 weeks. Intra- and subretinal fluid are assessed at each visit with optical coherence tomography (OCT). Should no intra- and subretinal fluid be present on OCT, the treatment interval to the next visit is extended by 2 weeks. Is intra- and or subretinal fluid present on OCT the treatment interval to the next visit is reduced by 2 weeks. The minimum treatment interval is 4 weeks, the maximum treatment interval is 12 weeks.
Number of injections received | during 32 weeks and 1 year
Proportion of eyes remaining on a 4-weekly interval from baseline to last visit (completed interval) | at 32 weeks and 56 weeks
  Treatment is administered at each visit. The interval between treatments is based on a treat and extend regime. The first interval between treatments, from baseline, is 4 weeks. Intra- and subretinal fluid are assessed at each visit with optical coherence tomography (OCT). Should no intra- and subretinal fluid be present on OCT, the treatment interval to the next visit is extended by 2 weeks. Is intra- and or subretinal fluid present on OCT the treatment interval to the next visit is reduced by 2 weeks. The minimum treatment interval is 4 weeks, the maximum treatment interval is 12 weeks.

OTHER OUTCOMES:
Mean change in ETDRS letter score | from baseline to an averaged EDTRS letter score between 24-32 weeks and between 48-56 weeks
  Best Corrected Visual Acuity (BCVA) is measured via Early Treatment Diabetic Retinopathy Severity (ETDRS) charts. The ETDRS letter score ranges from 0 to 100 (best score).
Mean averaged ETDRS letter score | between 24-32 weeks and between 48-56 weeks
  Best Corrected Visual Acuity (BCVA) is measured via Early Treatment Diabetic Retinopathy Severity (ETDRS) charts. The ETDRS letter score ranges from 0 to 100 (best score).
Proportion of eyes gaining ≥ 5 EDTRS letters | from baseline to an averaged ETDRS letter score between 24-32 weeks and between 48-56 weeks
Proportion of eyes loosing ≥5 EDTRS letters | from baseline to an averaged ETDRS letter score between 24-32 weeks and between 48-56 weeks
Mean change in low-luminance Best Corrected Visual Acuity (BCVA) | from baseline to last visit at or before 32 weeks and last visit at or before 56 weeks
Mean change in central subfield thickness (CST) | from baseline to an averaged CST between 24-32 weeks and between 48-56 weeks
  CST is measured using optical coherence tomography (OCT).
Proportion of eyes with no intraretinal fluid | at baseline, last visit at or before 32 weeks and at or before 56 weeks
  Intraretinal fluid is assessed via optical coherence tomography (OCT).
Proportion of eyes with no subretinal fluid | at baseline, last visit at or before 32 weeks and at or before 56 weeks
  Subretinal fluid is assessed via optical coherence tomography (OCT).
Proportion of eyes with no intra- and subretinal fluid | at baseline, last visit at or before 32 weeks and at or before 56 weeks
  Intra- and subretinal fluid is assessed via optical coherence tomography (OCT).
Retinal nerve fiber layer (RNFL) thickness | at baseline, last visit at or before 32 weeks and last visit at or before 56 weeks
  RNFL thickness is assessed via optical coherence tomography (OCT).
Concentration of plasma vascular endothelial growth factor A (VEGF-A) and Angiopoietin-2 (Ang-2) | at baseline, one week after baseline, four weeks after baseline and last visit at or before 32 weeks
  Plasma VEGF-A and Ang-2 is determined using a validated enzyme-linked immunosorbent assay (ELISA).
Patient-reported vision-related functioning and quality of life | at screening, last visit at or before 32 weeks and last visit at or before 56 weeks
  Patient-reported vision-related functioning and quality of life is assessed via National Eye Institute Visual Function Questionnaire (VFQ-25). VFQ-25 score ranges from 0 to 100 (highest score).
Presence of safety outcomes | from baseline through to week 56
  Rates of adverse events (AE's) and serious adverse events (SAE's) are given.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Wedrich, MD, Principal Investigator — Department of Ophthalmology, Medical University Graz
Locations (1):
- Department of Ophthalmolgy, Medical University Graz, Graz, Styria, Austria